CLINICAL TRIAL: NCT01136824
Title: Chemotherapy-induced Symptoms in Sarcoma Patients and the Impact of Tumor Burden
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 10-046
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma; questionnaire; doxorubicin plus ifosfamide (AI)
MeSH Terms: conditions — Sarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sarcoma Subjects: Soft tissue sarcoma patients treated with the adjuvant and neoadjuvant chemotherapy protocol of doxorubicin plus ifosfamide (AI)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Subjects will be given a series of questionnaires to assess the effect of AI chemotherapy, and the possible role of tumor load, on the amount of symptoms. The extent of nausea, vomiting, fatigue, anxiety, sleep disturbance, and cognitive changes will be measured. In adjuvant chemotherapy patients, we will also assess the relationship between tumor size and amount of chemotherapy-induced symptoms. These questionnaires will involve the following assessments:
  Demographic & health Trait anxiety Quality of life Nausea Expectations Anxiety & total mood disturbance Nausea & vomiting Multiple symptoms

SUMMARY:
Assessments (survey data) in this study are designed to sample the symptom burden of patients undergoing adjuvant and neoadjuvant chemotherapy in the hospital. There will be no change in the treatment plan for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving doxorubicin plus ifosfamide (AI)

Exclusion Criteria:

* There is no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Soft tissue sarcoma patients treated with the adjuvant and neoadjuvant chemotherapy protocol of doxorubicin plus ifosfamide (AI)
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine the extent of symptom burden and quality of life in sarcoma patients receiving AI chemotherapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, Principal Investigator — University of Pittsburgh; Charles Horn, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Hillman Cancer Center, Pittsburgh, Pennsylvania, United States